CLINICAL TRIAL: NCT03650439
Title: Fungal Infections In Patients With Hematological Malignancies In South Egypt Cancer Institute
Brief Title: Fungal Infections in Patients With Hematological Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Qwashty, Doctor, Assiut University
Other Study IDs: fungal infections
Record Dates: First submitted 2018-08-26; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: culture on Sabouraud's Dextrose Agar (SDA) — • Clinical samples will be cultured onto Sabouraud's Dextrose Agar (SDA) plates supplemented with chloramphenicol. the culture was incubated at 25 C° and at 37° C (for yeasts and moulds isolation )
  Other Names: E test

SUMMARY:
* Report the prevalence of fungal infections among patients with hematological malignancies in South Egypt Cancer Institute. * Detect the most endemic fungal pathogen isolated from patients with hematological malignancies in South Egypt Cancer Institute. *Antifungal susceptibility testing which guide the optimal approach to treat fungal infections. * detection of resistant gene expression by real time PCR. * Fungal genome sequencing analysis to determine the genetic back ground upon which mutation and resistance occur.

DETAILED DESCRIPTION:
Patients with hematologi¬cal malignancies are at increased risk of infections, not only because of the malignancy itself, but also because of neutropenia induced by intensive chemotherapy and its cyto¬toxic effect on the cells that line the gastrointestinal tract [1].

Invasive fungal infection (IFI) causes morbidity and mortality among patients with hematological malignancy.

The incidence of IFI has increased worldwide over the last two decades[2]. Major risk factors for IFI include neutropenia <500 neutrophils/ml for more than 10 days, bone marrow transplantation, prolonged (>4 wk) treatment with corticosteroids; prolonged (>7 days) stays in intensive care, chemotherapy, HIV infection, invasive medical procedures, and the newer immune suppressive agents. Other risk factors are malnutrition, solid organ transplantation, severe burns and major surgery [3].

Invasive aspergillosis (IA) and invasive candidiasis are the main invasive fungal diseases associated with bloodstream Infections. Although invasive yeasts, such as Candida spp., and molds, such as Aspergillus spp., are the predominant pathogens of IFIs, other uncommon and difficult-to-treat molds, such as Mucorales, Fusarium spp., and phaeohyphomycetes, have emerged in patients with hematological malignancies [4].

Early initiation of the correct antifungal therapy has been demonstrated to have a direct impact on the patient's outcome[5]. The increased use of antifungals has induced a higher selective pressure on fungal strains and resistance has emerged in two main ways: several species have developed secondary resistance and susceptible species have been replaced by resistant ones,changing the epidemiology of fungal infections[6]. Among the most common mechanisms of antifungal drug resistance are changes in the biosynthetic pathways targeted by drugs [7]. Genomics technology and the use of DNA microarrays have facilitated the identification of targets of novel antifungal drugs[8]. the molecular understanding of resistance mechanisms may identify fungal genes with mutations associated with resistance. Resistance mediated by alterations in Erg11/Cyp51 (targets of azoles) has been widely documented, involving either mutations or upregulation of their genes in Candida or Aspergillus species [9]. Up regulation of CDR1, CDR2, and MDR1 has been demonstrated in azole-resistant C. albicans [10]. Genome sequencing can type known drug resistance mutations , in some cases suggesting whether particular drugs will fail to control an infection .Whole genome variants could be screened for point mutations in specific drug targets that are highly correlated with resistance . for example , specific mutations in the target of azole drugs [11] .or in the transcription factors that control the expression of drug efflux transporters [12] can be identified from whole genome sequence data only in isolates that display drug resistance [13]. There are two general approaches for genomic analysis of fungal pathogens. One involves generation of a genome assembly de novo, such as for a species that has not been previously sequenced and assembled. In the other approach, commonly termed re-sequencing, variants are identified between an existing reference assembly and a sequenced isolate via alignment of sequence reads to the reference. However, the choice of technology selected to generate the sequence is influenced both by the approach selected and by the goals of the study .[14]

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised adult patient with hematological malignancy , risky to fungal infection as
* patients receiving cytotoxic or immunosuppressive therapy. Patients with prolonged and deep neutropenia.
* patients exposed to prolonged use of antibiotic , prolonged Foley catheter drainage peripheral I.V catheters, corticosteroid use
* patients have presentations of fungal infection such as pulmonary infections ( pneumonia , sinusitis). and disseminated infection manifested commonly as skin lesions or soft tissue involvement .

Exclusion Criteria:

* Non hematologicaly malignant patients .
* Any contraindication regarding procedure as:
* Local infection or distorted anatomy at the potential puncture site (eg, from previous surgical interventions,congenital or acquired malformations, or burns)
* Severe peripheral vascular disease of the limb involved

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study design that is intended to include adult patients with fungal infections as acomplication in hematologicayl malignant patients who would be recruited from South Egypt Cancer Institute outpatient clinic or inpatient ward
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
identification of endemic fungal pathogen in patients with hematological malignancies south Egypt cancer institute. | one year study
  Detect the most endemic fungal pathogen isolated from clinical sampels of patients with hematological malignancies in South Egypt Cancer Institute.